CLINICAL TRIAL: NCT06477770
Title: Granulated Sucrose as a Standard in Cesarean Section Surgical Wound Healing to Reduce Hospital Time. Single-blind Randomized Clinical Trial
Brief Title: Sucrose as a Standard in Cesarean Section Surgical Wound Healing to Reduce Hospital Time
Acronym: SAGRA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional Autonoma de Honduras (Other)
Responsible Party: Principal Investigator, Ricardo A Gutierrez Ramirez, MD, MSc, FACOG, Professor, research coordinator of the postgraduate course in gynecology and obstetrics, Universidad Nacional Autonoma de Honduras
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PGO-UNAH-47-2-2024
Record Dates: First submitted 2024-06-19; First posted 2024-06-27 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Surgical Wound Infection; Cesarean Wound; Dehiscence
MeSH Terms: conditions — Surgical Wound Infection | interventions — Sucrose

STUDY DESIGN:
Intervention Model Description: randomized, single-blind clinical trial, whose population to be studied will be randomized patients with a diagnosis of dehiscence and infection of a cesarean surgical wound who meet the inclusion and exclusion criteria.
Who Masked: Outcomes Assessor
Masking Description: Both the patients and 3 researchers will know the intervention, however, the groups will be listed and during the analysis phase, the analyst researcher will not know which group each patient corresponds to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The surgical wound will be washed with saline solution and 10 ml of chlorhexidine soap, then 75 g of sucrose will be administered to the surgical wound at 8:00 am every day, once a day, and then it will be covered with sterile gauze.
  Interventions: Procedure: Clorhexidine soap; Other: Sucrose
- Control (Sham Comparator): The surgical wound will be washed with saline solution and 10 ml of chlorhexidine soap, once a day, and then covered with sterile gauze.
  Interventions: Procedure: Clorhexidine soap

INTERVENTIONS:
Procedure: Clorhexidine soap — surgical wound will be washed with saline solution and 10 ml of chlorhexidine soap
Other: Sucrose — 75 g of sucrose will be administered to the surgical wound at 8:00 am every day, once a day, and then it will be covered with sterile gauze.
  Other Names: saccharose
  Arms: Intervention

SUMMARY:
It is a randomized, single-blind clinical trial, whose population to be studied will be randomized patients with a diagnosis of dehiscence and infection of a cesarean surgical wound who meet the inclusion and exclusion criteria.

H0: Sucrose does not reduce hospital days in patients with surgical wound dehiscence.

HA: Sucrose reduces hospital days in patients with surgical wound dehiscence.

DETAILED DESCRIPTION:
Cesarean section is one of the most performed surgical interventions at the Maternal and Child Hospital. Infection and dehiscence of the surgical site are some of the most common complications in post-cesarean section patients. The Honduran population, like those around the world, is susceptible to surgical site infections due to several risk factors and depends on each patient. Regarding the patients treated at the Maternal and Child Hospital, a surgical site risk of approximately 2-3% is estimated. Therefore, the investigators consider it beneficial to look for alternatives to treating surgical infections that help to reduce hospital time. Granulated sucrose has previously been used as a method for treating surgical wounds, however, no trial has been conducted to determine the benefits of its use.

Therefore, the investigators consider that it will be beneficial for the Gynecology and Obstetrics service of the Maternal and Child Hospital, especially the Septic ward, to carry out a study that helps to determine if the use of granulated sucrose reduces the hospitalization time of patients with infection and dehiscence of the surgical site due to cesarean section, as well as replacing the use of other methods that must be paid for by the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Delivery of a signed and dated informed consent form.
2. Declared willingness to comply with all study procedures and availability for the duration of the study.
3. Women from 18 to 45 years old
4. Enjoy good general health, as demonstrated by your medical history, and have been diagnosed with post-cesarean surgical wound dehiscence and fascia integra.
5. Ability to take oral medication and be willing to comply with the sucrose regimen.
6. Agreement to comply with Lifestyle Considerations

Exclusion Criteria:

1. Known allergic reactions to sucrose components.
2. Treatment with another investigational drug or other intervention within the previous 7 days.
3. Current smoker or tobacco consumption within the previous 3 months.
4. Treatment with antibiotics at least 2 weeks before hospitalization
5. Reinterventions before hospitalization

   -

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — puerperium
Enrollment: 24 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Changes of in-hospital days | from the first intervention to delayed primary closure (by third intention), on average less than 14 days
  from the intervention days

SECONDARY OUTCOMES:
Change of Satisfaction scale for scar assessment | 3 months
  Mesure with POSAS questionnaire (Patient and Observer Scar Assessment), The POSAS scale for the evaluation of scars is validated and shows advantages over other scales by integrating qualitative parameters and the opinion of the patient. It consists of six parameters to be evaluated on an ordinal scale from 1 to 10. The sum of all questions gives a final score (6 to 60 points). All items are rated on a scale ranging from 1 ("similar to normal skin") to 10 ("Very different from normal skin").
  Less points means a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo A. Gutierrez Ramirez, MD, MSc, Study Director — Universidad Nacional Autonoma de Honduras
Locations (1):
- Hospital Escuela, Tegucigalpa, Francisco Morazán Department, Honduras

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 12 months
Access Criteria: e mail

REFERENCES:
- [Background] Li S, Renick P, Senkowsky J, Nair A, Tang L. Diagnostics for Wound Infections. Adv Wound Care (New Rochelle). 2021 Jun;10(6):317-327. doi: 10.1089/wound.2019.1103. Epub 2020 Jul 7. PMID 32496977